CLINICAL TRIAL: NCT06444971
Title: Effects of Post-isometric Relaxation Technique on Chest Expansion and Pulmonary Function Tests in Smokers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/8
Record Dates: First submitted 2024-05-27; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: This study is a quasi pre test post test study with a single group. Participants will be recruited according to inclusion criteria .Each participant will receive same treatment .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PIR Group (Experimental): Post isometric relaxation technique will be applied to sternocleidomastoid and scalene muscles in all the participants with following parameters
  * Participant will perform isometric contractions using 20 -30% of their strength
  * HOLD TIME: 5-7 sec followed by 20 to 30 sec stretch
  * REST TIME: 5 sec
  * REPETITIONS: 3-5 repetitions
  Interventions: Procedure: Post isometric Relaxation

INTERVENTIONS:
Procedure: Post isometric Relaxation — Post isometric relaxation technique: It is defined as a manual procedure which involves the precisely controlled and specifically directed active contraction of a muscle at varying levels of intensity against a counterforce applied by the therapist.
  PIR will be applied to following muscles
  1. scalene (anterior, middle and posterior)
  2. sternocleidomastoid

SUMMARY:
The primary objective of the study was to investigate the immediate effects of PIR technique on chest expansion and pulmonary functions in cigarette smokers.This quasi-experimental pre-test post-test study will be conducted. Participants of interest would be approached and explained about the research. Informed written consent will be taken. Recruited participants will receive PIR technique on assessory respiratory muscles and chest expansion and pulmonary function tests will be obtained before and after the treatment. Data collection tools for this study are spirometer and measuring tape.

DETAILED DESCRIPTION:
Tobacco use, particularly cigarette smoking, is a major cause of disease and death globally. In Pakistan, the prevalence of tobacco use has increased significantly, with men being more likely to smoke than women. Chronic smoking is strongly associated with cardiovascular and respiratory diseases, as well as various forms of cancer. Smoking negatively affects lung function, leading to reduced pulmonary capacity and chronic obstructive pulmonary disease. Additionally, long-term smoking may lead to the loss of respiratory capacity and systemic muscle mass, affecting the performance and work of breathing.

The primary objective of the study was to investigate the effects of PIR technique on chest expansion and pulmonary functions in cigarette smokers.

This quasi-experimental pre-test post-test study will be conducted over one year at FFH, FUSH and among the general public. A sample will be calculated through pilot study. Participants between the ages of 18-60 will be recruited using convenience sampling. Inclusion criteria included individuals with min of 2 pack-years of tobacco smoking, while exclusion criteria included patients with certain cardiopulmonary medical conditions and those who underwent surgery or physiotherapy within past few months. Data collection tools for this study are spirometer and measuring tape.

There is little to no literature on the effects of PIR technique on chest expansion and pulmonary functions in cigarette smokers. The immediate effects of PIR technique demonstrated in this study will provide physical therapists with valuable insight into its use as a treatment option for smokers to improve their pulmonary function. Moreover, this study adds to the existing literature on manual therapy and its effects on smokers. The findings of this study will provide a basis for future research in the field of musculoskeletal rehabilitation and will encourage future researchers to explore this area further.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-60
* Only tobacco cigarette smokers
* Cigarette smokers (with min 2 pack years )
* Both males and females

Exclusion Criteria:

* Patients undergoing any surgery
* Symptomatic patients of cystic fibrosis, asthma, exercise induced asthma, unstable angina, bronchitis , bronchiectasis, chest deformities, congenital cardiopulmonary disorders , disc herniation, current rib or vertebral fracture
* Patients with a positive history of trauma, fracture or surgery of the cervical and thoracic spine in the last 12 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-06-25 (Estimated); Study Completion 2024-06-27 (Estimated)

PRIMARY OUTCOMES:
Chest expansion | Immediate after treatment
  Measuring tape will be used to measure chest expansion at axillary level.
Forced Vital Capacity(FVC) | Immediate after treatment
  the maximum amount of air you can forcibly exhale from your lungs after fully inhaling measured using hand held spirometer
Forced Expiratory Volume in 1 second (FEV1) | Immediate after treatment
  The volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration measured using hand held spirometer.
Peak Expiratory Flow (PEF) | Immediate after treatment
  the volume of air forcefully expelled from the lungs in one quick exhalation measured using hand held spirometer
FEV1/ FVC | Immediate after treatment
  The ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lung measured using hand held spirometer

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan